CLINICAL TRIAL: NCT01040065
Title: Distal Clavicle Resection of Symptomatic Acromioclavicular Joint Arthritis Combined With Rotator Cuff Tear. Prospective Randomized Trial
Brief Title: Distal Clavicle Resection With Rotator Cuff Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jae Chul Yoo, MD, Samsung Medical center
Other Study IDs: 2008-08-002
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Acromioclavicular Joint Arthritis
Keywords: Acromioclavicular joint arthritis; distal clavicle resection; Mumford procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: distal clavicle resection — Presence of tenderness at 2 years after surgery
  Other Names: mumford procedure

SUMMARY:
The purpose of this study is to determine whether distal clavicle resection is effective treatments in patients with acromioclavicular joint pain accompanied by rotator cuff tear.

DETAILED DESCRIPTION:
Today, acromioclavicular joint syndrome is itself rarely a cause for hospital visit, and the need for its treatment is even rarer. In comparison, patients who suffer rotator cuff tear accompanied by shoulder impingement syndrome often complain of acromioclavicular joint pain. However, often patients who complain of severe pain have no positive findings on X-ray or MRI, or any sign of impingement. On the other hand, there are patients with positive findings on X-ray or MRI who have only little pain. Even a patient who in the out-patient-department complained of acromioclavicular joint pain on pressure may feel pain on pressure in the physical exam performed for rotator cuff tear surgery. The opposite is very frequent as well, so it is often different depending on the time and the performer. In the literature, there are some authors who maintain that a distal clavicular resection must be done when surgery is used to treat the impingement syndrome, while on the other hand, there are those who endorse only complaining (an operation to trim the distal clavicle and the protruding part of adjust the plane acromion in order to level their plane), and also those who propose an all or none approach to either perform a distal clavicular resection or not at all. Thus, there are varying opinions depending on the authors; moreover, these are all observational studies, and none report on the rotator cuff tear injury. The authors of this study hypothesize and will prove that since the osteoarthritic change and pain of the acromioclavicular joint is secondary to impingement syndrome, distal clavicular resection on rotator cuff repair surgery will have no long term effect.

ELIGIBILITY:
Inclusion Criteria:

* rotator-cuff tear requiring repair
* acromioclavicular joint tenderness more than moderate(Pain Visual Analogue Scale 4-7)
* acromioclavicular arthritis(Petersson Grade II-III)

Exclusion Criteria:

* Arthritic changes of glenohumeral joint
* Combined infection
* Mini-open, open procedures
* Complete subscapularis tear
* Incomplete repair
* Neurologic abnormality including axillary nerve
* Adhesive capsulitis
* Prior surgery, trauma, or infection on shoulder girdle
* SLAP lesion or biceps tendon lesion without rotator-cuff tear or impingement syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medium sized rotator cuff tears
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
the presence of acromioclavicular joint tenderness | 2 years

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jae Chul Yoo, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Fischer BW, Gross RM, McCarthy JA, Arroyo JS. Incidence of acromioclavicular joint complications after arthroscopic subacromial decompression. Arthroscopy. 1999 Apr;15(3):241-8. doi: 10.1016/s0749-8063(99)70028-9. PMID 10231099
- [Result] Kharrazi FD, Busfield BT, Khorshad DS. Acromioclavicular joint reoperation after arthroscopic subacromial decompression with and without concomitant acromioclavicular surgery. Arthroscopy. 2007 Aug;23(8):804-8. doi: 10.1016/j.arthro.2007.02.003. PMID 17681199
- [Result] Kurta I, Datir S, Dove M, Rahmatalla A, Wynn-Jones C, Maffulli N. The short term effects of a single corticosteroid injection on the range of motion of the shoulder in patients with isolated acromioclavicular joint arthropathy. Acta Orthop Belg. 2005 Dec;71(6):656-61. PMID 16459853